CLINICAL TRIAL: NCT00001352
Title: Cryptococcosis in Previously Healthy Adults
Brief Title: Fungal Infection Susceptibility
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930106; 93-I-0106
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-10

CONDITIONS: Cryptococcal Infection; Cryptococcal Pneumonia; Pulmonary Cryptococcosis; Cryptococcal Meningitis; Cryptococcosis
Keywords: Natural History; Cryptococcus; Cryptococcus Neoformans; Cryptococcus gattii
MeSH Terms: conditions — Meningitis, Cryptococcal; Cryptococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Blood Relatives: Will be placed in a control group. Must be a blood relative of a patient enrolled in the study. Participant age must be 18 years or older. Relatives may be excluded if they have a condition that may interfere with evaluation of an immune system abnormality.
- Healthy Volunteers: Will be placed in a control group. Participant age must be 18 years or older. Healthy volunteers will be excluded if they have HIV, viral hepatitis (B or C), history of recurrent or severe infections, history of intravenous drug use, history of engaging in high-risk activities for HIV exposure, receiving chemotherapeutic agents, immunosuppressants, have underlying malignancies, pregnancy, or a history of heart disease, lung disease, kidney disease, or bleeding disorders.
- Patient Population: Previously healthy adult patients diagnosed with Cryptococcosis and have no predisposing conditions, such as HIV.

SUMMARY:
The protocol will be carried out in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) and the following United States Code of Federal Regulations (CFR) applicable to clinical studies: 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812.

NIH-funded investigators and study site staff who are responsible for the conduct, management, or oversight of NIH-funded studies have completed Human Subjects Protection and ICH GCP Training.

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be approved by the IRB; an IRB determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

...

DETAILED DESCRIPTION:
Cryptococcus is a fungus that causes infections most commonly in immunocompromised patients, such as those with AIDS and solid organ transplant recipients, particularly renal transplant recipients (1-3). However, approximately one-third of cases fall outside these groups and, overall, 12.9 percent to 17.9 percent have no readily identifiable immune defect (4, 5). The genetic factors, which may predispose to cryptococcosis and the immune response in these patients, have not been extensively studied.

This protocol is designed to examine the immune deficits that predispose to cryptococcosis as well as the clinical and immune responses among previously healthy adults. The patients included will have an unknown predisposing condition and cryptococcosis. Patients will undergo various sampling procedures, including saliva, blood, eyebrow hair, CSF, and nail clipping collection. Throughout the study, patients will be provided with standard medical care and will be seen as often as necessary to manage their condition. Patients in whom microbiologic control of the infection has occurred but in whom inflammation is causing neurologic damage may be treated with corticosteroids or other immunosuppressive agents. Genetically related family members of patients will also be screened for clinical, in vitro, immune, and genetic correlates of immune abnormalities. Healthy adult volunteers, as a comparison group, will be enrolled as a source of blood samples, saliva samples, CSF samples, and eyebrow hair samples for research testing. Moreover, with respect to cryptococcosis, patients with isolated non-central nervous system (CNS) disease (e.g., pulmonary) may serve as a subset comparator to those with CNS involvement-a major tissue tropism for Cryptococcus.

Genetic and immunologic testing will be performed on all subjects (patients, relatives, and healthy volunteers) to evaluate for possible immunogenetic factors that lead to susceptibility to cryptococcosis. Among the aims of this protocol are to better understand the pathophysiology and genetic factors that lead to defects in host defense and to use modern and evolving methods in molecular and cellular biology to elucidate the pathogenesis of this particular susceptibility. A better understanding of the underlying pathophysiology of immune defects and genetic susceptibility to fungal infections could allow for the rational development of novel therapies for such diseases and to benefit future patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients

Patients must:

1. Have cryptococcosis as determined by information collected from their medical records, telephone interviews, or from a referring physician:

   * histopathology showing cryptococci; or
   * culture of C. neoformans or C. gattii
   * a positive cryptococcal antigen in the serum and/or CSF, together with CSF cell count and chemistry consistent with cryptococcal meningitis.
2. Be over the age of 18 years old.
3. Have a primary physician outside of the NIH.
4. Agree to undergo genetic testing that will include WES and high density SNP arrays as appropriate for possible WES linkage studies.
5. Allow samples to be stored for future research.
6. Pregnant patients will not be excluded. However, research procedures greater than minimal risk including bone marrow biopsy and apheresis would not be performed on pregnant subjects. Otherwise, pregnant patients with cryptococcus would be treated with as per standard of care, minimizing teratogenic potential of drugs and ionizing radiation whenever possible.

Blood Relatives of Patients

Blood relatives must:

1. Be a genetic relative of a patient enrolled in this study
2. Be over the age of 18 years old
3. Agree to undergo genetic testing that may include WES and high density SNP analysis
4. Allow samples to be stored for future research

Healthy Volunteers

Healthy volunteers must:

1. Be between the ages of 18 and 70 years old
2. Allow samples to be stored for future research

EXCLUSION CRITERIA:

Patients

Patients will be excluded for any of the following:

1. The presence of certain types of acquired abnormalities of immunity due to:

   * HIV
   * Cancer chemotherapeutic agent(s)
   * An underlying malignancy could be grounds for possible exclusion of a patient if, in the opinion of the investigator, the underlying disease predisposed the patient to the infection
   * Monoclonal antibody therapy directed against a patient s immune system
2. Any condition that in the opinion of the investigator may interfere with the evaluation of a co-existing abnormality of immunity that is the subject of study under this protocol. For example, we may exclude patients with Cushing s disease that have very high cortisol levels at the time of diagnosis of their cryptococcosis.

Genetic Relatives of Patients

Genetic relatives will be excluded for the following:

-Any condition that in the opinion of the investigator may interfere with evaluation of an immune system abnormality that is the subject of study under this protocol.

Healthy Volunteers

Healthy volunteers will be excluded for any of the following:

1. HIV or viral hepatitis (B or C).
2. History of recurrent or severe infections.
3. History of intravenous drug use.
4. History of engaging in high-risk activities for exposure to HIV.
5. Receiving chemotherapeutic agent(s), immunosuppressants or have underlying malignancy.
6. Pregnancy.
7. Have history of heart, lung, kidney disease, or bleeding disorders.
8. Any condition that in the opinion of the investigator may interfere with evaluation of an immune system abnormality that is the subject of study under this protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will consist of previously healthy adults without known prior conditions who have cryptococcosis, blood relatives of these patients, and healthy adult volunteers. Potential Cryptococcus patients must be 18 or older with evidence of positive Cryptococcus infection results as shown through their medical records, telephone interviews or referring physician. This includes a positive Cryptococcus culture (neoformans or gattii), a positive cryptococcal antigen from serum or CSF with CSF cell count and chemistry consistent with Cryptococcus infection, or histopathology showing cryptococci. Blood relatives and healthy volunteers must be 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1993-04-01 (Actual)

PRIMARY OUTCOMES:
Characterize the full spectrum of clinical disease of Cryptococcosis in previously healthy adults without known immune predisposition. | 1-5 years

SECONDARY OUTCOMES:
Characterize the immunological and genetic mechanisms predisposing to disease acquisition. | 1-5 years
Understand the inflammatory response and distinguish its consequences from those directly due to fungal growth. | 1-5 years
Understand the natural history of disease progression or regression over time. | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Williamson, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baddley JW, Forrest GN; AST Infectious Diseases Community of Practice. Cryptococcosis in solid organ transplantation. Am J Transplant. 2013 Mar;13 Suppl 4:242-9. doi: 10.1111/ajt.12116. No abstract available. PMID 23465017
- [Background] Park BJ, Wannemuehler KA, Marston BJ, Govender N, Pappas PG, Chiller TM. Estimation of the current global burden of cryptococcal meningitis among persons living with HIV/AIDS. AIDS. 2009 Feb 20;23(4):525-30. doi: 10.1097/QAD.0b013e328322ffac. PMID 19182676
- [Background] Perfect JR, Dismukes WE, Dromer F, Goldman DL, Graybill JR, Hamill RJ, Harrison TS, Larsen RA, Lortholary O, Nguyen MH, Pappas PG, Powderly WG, Singh N, Sobel JD, Sorrell TC. Clinical practice guidelines for the management of cryptococcal disease: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2010 Feb 1;50(3):291-322. doi: 10.1086/649858. PMID 20047480
- [Background] Brizendine KD, Baddley JW, Pappas PG. Predictors of mortality and differences in clinical features among patients with Cryptococcosis according to immune status. PLoS One. 2013;8(3):e60431. doi: 10.1371/journal.pone.0060431. Epub 2013 Mar 26. PMID 23555970
- [Background] Bratton EW, El Husseini N, Chastain CA, Lee MS, Poole C, Sturmer T, Juliano JJ, Weber DJ, Perfect JR. Comparison and temporal trends of three groups with cryptococcosis: HIV-infected, solid organ transplant, and HIV-negative/non-transplant. PLoS One. 2012;7(8):e43582. doi: 10.1371/journal.pone.0043582. Epub 2012 Aug 24. PMID 22937064
- [Background] Gullo FP, Rossi SA, Sardi Jde C, Teodoro VL, Mendes-Giannini MJ, Fusco-Almeida AM. Cryptococcosis: epidemiology, fungal resistance, and new alternatives for treatment. Eur J Clin Microbiol Infect Dis. 2013 Nov;32(11):1377-91. doi: 10.1007/s10096-013-1915-8. Epub 2013 Jul 4. PMID 24141976
- [Background] Baddley JW, Perfect JR, Oster RA, Larsen RA, Pankey GA, Henderson H, Haas DW, Kauffman CA, Patel R, Zaas AK, Pappas PG. Pulmonary cryptococcosis in patients without HIV infection: factors associated with disseminated disease. Eur J Clin Microbiol Infect Dis. 2008 Oct;27(10):937-43. doi: 10.1007/s10096-008-0529-z. Epub 2008 May 1. PMID 18449582
- [Background] Chen SC, Korman TM, Slavin MA, Marriott D, Byth K, Bak N, Currie BJ, Hajkowicz K, Heath CH, Kidd S, McBride WJ, Meyer W, Murray R, Playford EG, Sorrell TC; Australia and New Zealand Mycoses Interest Group (ANZMIG) Cryptococcus Study. Antifungal therapy and management of complications of cryptococcosis due to Cryptococcus gattii. Clin Infect Dis. 2013 Aug;57(4):543-51. doi: 10.1093/cid/cit341. Epub 2013 May 22. PMID 23697747
- [Background] Pappas PG. Cryptococcal infections in non-HIV-infected patients. Trans Am Clin Climatol Assoc. 2013;124:61-79. PMID 23874010
- [Background] Meletiadis J, Walsh TJ, Choi EH, Pappas PG, Ennis D, Douglas J, Pankey GA, Larsen RA, Hamill RJ, Chanock S. Study of common functional genetic polymorphisms of FCGR2A, 3A and 3B genes and the risk for cryptococcosis in HIV-uninfected patients. Med Mycol. 2007 Sep;45(6):513-8. doi: 10.1080/13693780701390140. PMID 17710620
- [Background] Schepelmann K, Muller F, Dichgans J. Cryptococcal meningitis with severe visual and hearing loss and radiculopathy in a patient without immunodeficiency. Mycoses. 1993 Nov-Dec;36(11-12):429-32. doi: 10.1111/j.1439-0507.1993.tb00734.x. PMID 7935577
- [Background] Rosen LB, Freeman AF, Yang LM, Jutivorakool K, Olivier KN, Angkasekwinai N, Suputtamongkol Y, Bennett JE, Pyrgos V, Williamson PR, Ding L, Holland SM, Browne SK. Anti-GM-CSF autoantibodies in patients with cryptococcal meningitis. J Immunol. 2013 Apr 15;190(8):3959-66. doi: 10.4049/jimmunol.1202526. Epub 2013 Mar 18. PMID 23509356
- [Background] Rabbani B, Tekin M, Mahdieh N. The promise of whole-exome sequencing in medical genetics. J Hum Genet. 2014 Jan;59(1):5-15. doi: 10.1038/jhg.2013.114. Epub 2013 Nov 7. PMID 24196381
- [Background] Mullaney JM, Mills RE, Pittard WS, Devine SE. Small insertions and deletions (INDELs) in human genomes. Hum Mol Genet. 2010 Oct 15;19(R2):R131-6. doi: 10.1093/hmg/ddq400. Epub 2010 Sep 21. PMID 20858594
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1993-I-0106.html